CLINICAL TRIAL: NCT00259454
Title: Managing Problem Behaviors of Alzheimer's Disease
Brief Title: Project COPE:Managing Dementia at Home
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Laura N. Gitlin, Ph.D, Thomas Jefferson Univeristy-Center for Applied Research on Aging and Health
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SAP 4100027298
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Dementia, Alzheimer Type
Keywords: Caregivers; in-home care occupational therapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: In-home intervention — occupational therapy techniques to reduce caregiver stress

SUMMARY:
This study tests the effectiveness of an in-home intervention to reduce upset and burden among family caregivers, and decrease nursing home placement. The main hypothesis that will be tested is that compared to control group, subjects, experimental group participants will have enhanced well-being and fewer nursing home placements.

DETAILED DESCRIPTION:
Implement a multi-component in-home intervention designed to prevent and ameliorate the troublesome behaviors that families typically confront and that often trigger nursing home placement. The intervention combines the most effective strategies that have been identified in previous caregiver research by the investigative team and best clinical practices to provide a comprehensive service approach to families and individuals with dementia including education, skills training, home safety, and stress management. To enhance its applicability to real-world practice within the aging service network, the intervention is designed to be reproducible and its components and treatment goals commensurate with the Medicaid Waiver Program. In the absence of evidence-based service protocols currently in place for this Waiver population, the intervention, if effective, would provide a systematic, evidence-based approach in the Medicaid Waiver program to help families and persons with dementia remain at home and in their communities.

ELIGIBILITY:
Inclusion Criteria:

* Care-recipients must have a MMSE score < 24 and a diagnosis of dementia, live in the community, and either need help with one or more daily activities and/or have one or more behavioral occurrences. Caregivers must be a relative, at least 21 years of age, be English speaking, have a telephone, either live with the care-recipient (CR) or spend at least 48 hours per week in direct oversight or caring for him/her; plan to live in the area for 9 months, report upset with CR function dependence or behavioral occurrences.

Exclusion Criteria:

* The CG-CR dyad will be excluded if CR has had more than 3 hospitalizations within the past 12 months, are in treatment for life-threatening cancer, have schizophrenia or a bipolar disorder, have dementia secondary to head trauma, have a MMSE score = 0 and are bed-bound (defined as confinement to bed or chair for at least 22 hours a day for at least four of the previous seven days); or they are enrolled in a clinical trial of pharmacological treatment for agitation. Also, the dyad will be excluded if the CG had more than 3 hospitalizations within the past 12 months or is in treatment for life-threatening cancer; is involved in another clinical trial of psychosocial or educational interventions for caregivers; or plans to place their family member in a nursing home within the next 9-months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
ADL/IADL | Baseline, t2, t3
Caregiver upset | Baseline, t2, t3
Caregiver confidence | when needed
Behaviors | Baseline, t2, t3

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, Ph.D, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Hodgson NA, Gitlin LN, Winter L, Czekanski K. Undiagnosed illness and neuropsychiatric behaviors in community residing older adults with dementia. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):109-15. doi: 10.1097/WAD.0b013e3181f8520a. PMID 20921879
- [Derived] Gitlin LN, Winter L, Dennis MP, Hodgson N, Hauck WW. A biobehavioral home-based intervention and the well-being of patients with dementia and their caregivers: the COPE randomized trial. JAMA. 2010 Sep 1;304(9):983-91. doi: 10.1001/jama.2010.1253. PMID 20810376
- See also: Farber Institute for Neurosciences of Thomas Jefferson University — http://www.jefferson.edu/fin/